CLINICAL TRIAL: NCT03554915
Title: Ketamine Versus Midazolam for Prehospital Agitation
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HSR #17-4306
Record Dates: First submitted 2018-05-29; First posted 2018-06-13 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Agitation
Keywords: Agitation, Ketamine, Midazolam, Emergency Medical Services
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ketamine-based Protocol: The first 6 month period of the study will employ a ketamine-based protocol for prehospital agitation. There will be a tiered dosing protocol based on degree of agitation.
  Interventions: Other: Ketamine-based protocol
- Midazolam-based Protocol: The second 6 month period of the study will employ a midazolam-based protocol for prehospital agitation. There will again be a tiered dosing protocol based on degree of agitation.
  Interventions: Other: Midazolam-based protocol

INTERVENTIONS:
Other: Ketamine-based protocol — For profoundly agitated (physically violent) patients, intramuscular ketamine 5 mg/kg will be administered first line. For severely agitated patients, intramuscular ketamine 3 mg/kg will be administered first line.
  Groups: Ketamine-based Protocol
Other: Midazolam-based protocol — For profoundly agitated patients, intramuscular midazolam 15 mg will be administered. For severely agitated patients, intramuscular midazolam 5 mg will be administered.
  Groups: Midazolam-based Protocol

SUMMARY:
This research study is being done to figure out the best approach to treatment of pre-hospital agitation. It will compare two tiered dosing treatment protocols, one ketamine-based and one midazolam-based. Agitation is a state of extreme emotional disturbance where patients can become physically aggressive or violent, endangering themselves and those who are caring for them. Often chemical substances or severe mental illness are involved in this level of agitation. Specifically, the investigators are interested in studying agitation that is treated in the prehospital setting by paramedics. This study's hypothesis is a ketamine-based protocol will achieve a faster time to adequate sedation than a midazolam-based protocol for treatment of agitation in the prehospital environment. This study will observe the natural history of an emergency medical services standard operating procedure change from a ketamine-based protocol to a midazolam-based protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Severe agitation (AMSS +2 or +3) or profound agitation (AMSS +4) requiring chemical sedation
* Transport to Hennepin County Medical Center

Exclusion Criteria:

* Obviously gravid women
* Patients known or suspected to be less than 18 years of age
* Patients in which stopwatch activation, for safety reasons, is unable to occur

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is all patients over age 18 requiring chemical sedation for transport to the emergency department. Etiologies for agitation may include mental illness, substance abuse, critical illness or undetermined.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Time from injection of drug to adequate sedation, defined as a score of +1 or less on the AMSS | 2 hours
  The Altered Mental Status Scale (AMSS) is an integral ordinal scale evaluating both agitation and sedation with scores from -4 to +4. It was developed at our institution and has been internally and externally validated. This scale is a modified version of the Behavioral Activity Rating Scale with additional data points from the Observer's Assessment of Alertness Scale. Effectiveness of sedation will be defined as an AMSS score less than or equal to +1.
  AMSS will be determined by the treating paramedic, who will undergo training as a research associate prior to commencement of the study. Participants will be followed for the duration of agitation, an expected average of 2 hours.

SECONDARY OUTCOMES:
Number of participants intubated | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if the patient is intubated.
Number of participants experiencing hypersalivation | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if the patient experiences hypersalivation.
Number of participants experiencing apnea | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if the patient experiences apnea, defined as 6 seconds of absent EtCO2 waveform.
Number of participants experiencing nausea/vomiting | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if the patient experiences nausea/vomiting
Number of participants experiencing laryngospasm | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if laryngospasm occurs.
Number of participants needing rescue sedation | 2 hours
  Participants will be followed for the duration of agitation, an expected average of 2 hours. Enrolling paramedics or research associates in the Emergency Department will record if additional sedatives are needed in the prehospital or ED environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole JB, Klein LR, Nystrom PC, Moore JC, Driver BE, Fryza BJ, Harrington J, Ho JD. A prospective study of ketamine as primary therapy for prehospital profound agitation. Am J Emerg Med. 2018 May;36(5):789-796. doi: 10.1016/j.ajem.2017.10.022. Epub 2017 Oct 7. PMID 29033344
- [Background] Olives TD, Nystrom PC, Cole JB, Dodd KW, Ho JD. Intubation of Profoundly Agitated Patients Treated with Prehospital Ketamine. Prehosp Disaster Med. 2016 Dec;31(6):593-602. doi: 10.1017/S1049023X16000819. Epub 2016 Sep 19. PMID 27640730
- [Background] Cole JB, Moore JC, Nystrom PC, Orozco BS, Stellpflug SJ, Kornas RL, Fryza BJ, Steinberg LW, O'Brien-Lambert A, Bache-Wiig P, Engebretsen KM, Ho JD. A prospective study of ketamine versus haloperidol for severe prehospital agitation. Clin Toxicol (Phila). 2016 Aug;54(7):556-62. doi: 10.1080/15563650.2016.1177652. Epub 2016 Apr 22. PMID 27102743
- [Background] Ho JD, Smith SW, Nystrom PC, Dawes DM, Orozco BS, Cole JB, Heegaard WG. Successful management of excited delirium syndrome with prehospital ketamine: two case examples. Prehosp Emerg Care. 2013 Apr-Jun;17(2):274-9. doi: 10.3109/10903127.2012.729129. Epub 2012 Dec 11. PMID 23231451
- [Background] TREC Collaborative Group. Rapid tranquillisation for agitated patients in emergency psychiatric rooms: a randomised trial of midazolam versus haloperidol plus promethazine. BMJ. 2003 Sep 27;327(7417):708-13. doi: 10.1136/bmj.327.7417.708. PMID 14512476
- [Background] Page CB, Parker LE, Rashford SJ, Bosley E, Isoardi KZ, Williamson FE, Isbister GK. A Prospective Before and After Study of Droperidol for Prehospital Acute Behavioral Disturbance. Prehosp Emerg Care. 2018 Nov-Dec;22(6):713-721. doi: 10.1080/10903127.2018.1445329. Epub 2018 Mar 20. PMID 29558224
- [Background] Isbister GK, Calver LA, Page CB, Stokes B, Bryant JL, Downes MA. Randomized controlled trial of intramuscular droperidol versus midazolam for violence and acute behavioral disturbance: the DORM study. Ann Emerg Med. 2010 Oct;56(4):392-401.e1. doi: 10.1016/j.annemergmed.2010.05.037. PMID 20868907
- [Background] Scaggs TR, Glass DM, Hutchcraft MG, Weir WB. Prehospital Ketamine is a Safe and Effective Treatment for Excited Delirium in a Community Hospital Based EMS System. Prehosp Disaster Med. 2016 Oct;31(5):563-9. doi: 10.1017/S1049023X16000662. Epub 2016 Aug 12. PMID 27517801
- [Background] Martel M, Miner J, Fringer R, Sufka K, Miamen A, Ho J, Clinton J, Biros M. Discontinuation of droperidol for the control of acutely agitated out-of-hospital patients. Prehosp Emerg Care. 2005 Jan-Mar;9(1):44-8. doi: 10.1080/10903120590891723. PMID 16036827
- [Background] Keseg D, Cortez E, Rund D, Caterino J. The Use of Prehospital Ketamine for Control of Agitation in a Metropolitan Firefighter-based EMS System. Prehosp Emerg Care. 2015 January-March;19(1):110-115. doi: 10.3109/10903127.2014.942478. Epub 2014 Aug 25. PMID 25153713
- [Background] Hollis GJ, Keene TM, Ardlie RM, Caldicott DG, Stapleton SG. Prehospital ketamine use by paramedics in the Australian Capital Territory: A 12 month retrospective analysis. Emerg Med Australas. 2017 Feb;29(1):89-95. doi: 10.1111/1742-6723.12685. Epub 2016 Oct 3. PMID 27699989
- [Background] Isenberg DL, Jacobs D. Prehospital Agitation and Sedation Trial (PhAST): A Randomized Control Trial of Intramuscular Haloperidol versus Intramuscular Midazolam for the Sedation of the Agitated or Violent Patient in the Prehospital Environment. Prehosp Disaster Med. 2015 Oct;30(5):491-5. doi: 10.1017/S1049023X15004999. Epub 2015 Sep 1. PMID 26323511
- [Background] Scheppke KA, Braghiroli J, Shalaby M, Chait R. Prehospital use of i.m. ketamine for sedation of violent and agitated patients. West J Emerg Med. 2014 Nov;15(7):736-41. doi: 10.5811/westjem.2014.9.23229. Epub 2014 Nov 11. PMID 25493111
- [Background] Cole JB, Driver BE, Klein LR, Moore JC, Nystrom PC, Ho JD. In reply: Ketamine is an important therapy for prehospital agitation - Its exact role and side effect profile are still undefined. Am J Emerg Med. 2018 Mar;36(3):502-503. doi: 10.1016/j.ajem.2017.12.014. Epub 2017 Dec 7. No abstract available. PMID 29229535
- [Background] Linder LM, Ross CA, Weant KA. Ketamine for the Acute Management of Excited Delirium and Agitation in the Prehospital Setting. Pharmacotherapy. 2018 Jan;38(1):139-151. doi: 10.1002/phar.2060. Epub 2017 Dec 22. PMID 29136301
- [Background] Parsch CS, Boonstra A, Teubner D, Emmerton W, McKenny B, Ellis DY. Ketamine reduces the need for intubation in patients with acute severe mental illness and agitation requiring transport to definitive care: An observational study. Emerg Med Australas. 2017 Jun;29(3):291-296. doi: 10.1111/1742-6723.12763. Epub 2017 Mar 20. PMID 28320079
- [Background] Miner JR. Ketamine is a good first-line option for severely agitated patients in the prehospital environment. Am J Emerg Med. 2018 Mar;36(3):501-502. doi: 10.1016/j.ajem.2017.12.015. Epub 2017 Dec 7. No abstract available. PMID 29329930
- [Background] Buckland DM, Crowe RP, Cash RE, Gondek S, Maluso P, Sirajuddin S, Smith ER, Dangerfield P, Shapiro G, Wanka C, Panchal AR, Sarani B. Ketamine in the Prehospital Environment: A National Survey of Paramedics in the United States. Prehosp Disaster Med. 2018 Feb;33(1):23-28. doi: 10.1017/S1049023X17007142. Epub 2017 Dec 21. PMID 29265995
- [Background] Gonin P, Beysard N, Yersin B, Carron PN. Excited Delirium: A Systematic Review. Acad Emerg Med. 2018 May;25(5):552-565. doi: 10.1111/acem.13330. Epub 2017 Nov 27. PMID 28990246
- [Background] Melamed E, Oron Y, Ben-Avraham R, Blumenfeld A, Lin G. The combative multitrauma patient: a protocol for prehospital management. Eur J Emerg Med. 2007 Oct;14(5):265-8. doi: 10.1097/MEJ.0b013e32823a3c9b. PMID 17823561
- [Background] Cong ML, Humble I. A Ketamine Protocol and Intubation Rates for Psychiatric Air Medical Retrieval. Air Med J. 2015 Nov-Dec;34(6):357-9. doi: 10.1016/j.amj.2015.07.007. PMID 26611223
- [Background] Hick JL, Ho JD. Ketamine chemical restraint to facilitate rescue of a combative "jumper". Prehosp Emerg Care. 2005 Jan-Mar;9(1):85-9. doi: 10.1080/10903120590891859. No abstract available. PMID 16036834
- [Background] Burnett AM, Peterson BK, Stellpflug SJ, Engebretsen KM, Glasrud KJ, Marks J, Frascone RJ. The association between ketamine given for prehospital chemical restraint with intubation and hospital admission. Am J Emerg Med. 2015 Jan;33(1):76-9. doi: 10.1016/j.ajem.2014.10.016. Epub 2014 Oct 22. PMID 25455046
- [Background] Martel M, Sterzinger A, Miner J, Clinton J, Biros M. Management of acute undifferentiated agitation in the emergency department: a randomized double-blind trial of droperidol, ziprasidone, and midazolam. Acad Emerg Med. 2005 Dec;12(12):1167-72. doi: 10.1197/j.aem.2005.07.017. Epub 2005 Nov 10. PMID 16282517